CLINICAL TRIAL: NCT07274358
Title: HopeMove: Feasibility and Acceptability of a Mobile Application to Promote Physical Activity in Pediatric Hemotology and Oncology Patients
Brief Title: HopeMove App in Pediatric Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Koç University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Eysan Hanzade Umac, Teaching and Research Assistant, Koç University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: KOCUN
Record Dates: First submitted 2025-11-27; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Physical Activity; Mobile Application
Keywords: physical activity, fatigue, quality of life, mobile application
MeSH Terms: conditions — Motor Activity; Fatigue

STUDY DESIGN:
Intervention Model Description: Single-arm pilot feasibility study in which all participants receive the HopeMove intervention without a comparison group.
Masking Description: Masking was not applied due to the nature of the intervention, and all participants and investigators were aware of the intervention being delivered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group-HopeMove Application Group (Experimental): Participants assigned to the HopeMove Application Group will use HopeMove, a mobile application designed to promote and support physical activity among pediatric hematology and oncology patients. During the 4-week feasibility period, participants are instructed to engage with the application at least 3 days per week, completing the guided physical activity sessions provided within the app.
  Interventions: Other: HopeMove Mobile Application

INTERVENTIONS:
Other: HopeMove Mobile Application — HopeMove is a mobile application developed to promote physical activity and support wellbeing among pediatric hematology-oncology patients. The application provides age-appropriate guided exercise sessions, motivational prompts, visual progress tracking, and individualized activity suggestions tailored to each participant's needs and abilities.
  During the feasibility study, participants were instructed to engage with the HopeMove application at least three days per week for a total duration of four weeks. Each session included structured physical activity modules designed to be safe and achievable during hospitalization or home recovery.
  The intervention focused on feasibility, usability, acceptability, and preliminary effects on outcomes such as fatigue and satisfaction. No masking was applied due to the nature of the digital intervention.

SUMMARY:
This pilot feasibility study aims to assess the acceptability, usability, safety, and initial effects of the HopeMove mobile health app on fatigue in adolescents aged 13 to 18 years undergoing hematology-oncology treatment. HopeMove is a wearable-compatible app that offers guided home exercise sessions and daily symptom tracking to support physical activity and monitor well-being during treatment. The study includes an expert usability evaluation with 10 clinicians, a one-week usability testing phase with 15 adolescents, and an eight-week intervention period in which participants complete at least three exercise sessions per week using the app. Outcomes include usability measured with the Mobile Application Usability Scale, satisfaction assessed via a Visual Analog Scale, and fatigue evaluated with the Fatigue Scale. The findings are expected to provide evidence on the feasibility, usability, and potential clinical benefits of mobile-supported exercise programs for children and adolescents undergoing cancer treatment.

DETAILED DESCRIPTION:
Adolescents undergoing cancer treatment often face declines in physical function, decreased physical activity, and cancer-related fatigue, all of which negatively impact their quality of life and treatment adherence. Reduced activity and extended hospital stays can worsen fatigue and emotional distress, limiting daily activities and overall well-being. Exercise-based supportive care programs have proven beneficial in pediatric oncology, but access to structured, developmentally suitable options remains limited. Mobile health solutions are emerging as a way to support physical activity and symptom monitoring through accessible digital platforms.

HopeMove is a mobile app designed to encourage physical activity and symptom tracking among adolescents aged 13-18 years receiving hematology-oncology treatment. The app features short guided exercise videos, daily symptom diaries, weekly activity summaries, and compatibility with wearable devices.

The evaluation was carried out in three successive phases. First, 10 clinical experts reviewed the app using the Mobile Application Usability Scale to evaluate clarity, usability, and clinical appropriateness. Next, 15 adolescents participated in a one-week usability test, during which they used the app and provided structured feedback. In addition to quantitative usability scores, adolescents completed an 8-item open-ended interview developed by the research team to assess ease of use, clarity of instructions, comfort during exercise, content relevance, and expectations. Feedback from experts and adolescents was combined to improve the app before proceeding.

In the third phase, the same 15 adolescents used HopeMove over eight weeks. They were instructed to complete at least three guided exercise sessions weekly, with the option for additional sessions. During the intervention, adolescents also performed daily in-app symptom check-ins responding to "How do you feel today?" with a visual rating scale to record their overall perceived condition each day. Fatigue was measured at baseline and after the intervention using the Fatigue Scale, and satisfaction was assessed with a Visual Analog Scale. Adherence, usability, and safety were monitored throughout, with no adverse events reported.

This pilot feasibility study aims to assess the usability, acceptability, safety, and preliminary clinical effects of the HopeMove app in adolescents receiving hematology-oncology treatment. Results are expected to provide evidence supporting the potential benefits of mobile app-based exercise interventions for children and adolescents undergoing cancer treatment and to inform the design of future controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* adolescents aged 13-18 years
* receiving active hematology-oncology treatment
* able to use a smartphone running Android operating system
* has internet access
* voluntarily agrees to participate
* parent/guardian consent obtained (if applicable)
* able to perform light-moderate exercise
* able to complete at least 75% of planned exercise sessions

Exclusion Criteria:

* having a chronic illness requiring regular invasive procedures,
* having received analgesics within the past 2 hours,
* having experienced a seizure within the past 2 hours,
* using antiepileptic medication,
* having a body temperature above 37.5°C
* not having parental consent,
* being agitated at the time of the procedure,
* having any auditory or visual impairments.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2025-08-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Mobile Application Usability | Prior to the initiation of the pilot trial (single assessment during the development phase)
  Mobile application usability was evaluated prior to the pilot study by a panel of experts in pediatric oncology, digital health, and user-centered design. Experts assessed the HopeMove application using a standardized usability assessment form that examined clarity of content, ease of navigation, appropriateness for the target age group, visual design, responsiveness, and overall user experience. Feedback from experts was used to refine and optimize the application before initiating the pilot trial.
Fatigue | Baseline (initial meeting) and Week 4 (end of feasibility period)
  Fatigue levels were assessed to evaluate the preliminary effectiveness of the HopeMove mobile application. Fatigue was measured using a standardized pediatric fatigue assessment tool administered before the intervention (at the initial meeting) and at the end of the 4-week feasibility period. Changes in fatigue scores were examined to explore whether engagement with the application was associated with improvements in perceived fatigue among participants.

SECONDARY OUTCOMES:
Satisfaction for Mobile Application | Week 4 (end of feasibility period)
  Participant satisfaction with the HopeMove mobile application was evaluated to assess overall acceptability of the intervention. Satisfaction was measured using a structured satisfaction questionnaire administered at the end of the 4-week feasibility period. The questionnaire assessed perceived usefulness, enjoyment, clarity of instructions, willingness to continue using the app, and overall satisfaction. Higher scores indicated greater satisfaction with the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains identifiable health information of pediatric participants, and sharing is restricted to protect patient privacy in accordance with ethical and legal requirements.